CLINICAL TRIAL: NCT00654433
Title: A Phase III Trial of ALD-101 Adjuvant Therapy of Unrelated Umbilical Cord Blood Transplantation (UCBT) in Patients With Inborn Errors of Metabolism
Brief Title: ALD-101 Adjuvant Therapy of Unrelated Umbilical Cord Blood Transfusion (UCBT) in Patients With Inherited Metabolic Diseases
Acronym: UCBT-002
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated - Sponsor Decision
Sponsor: Aldagen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBT-002; BB-IND#13502
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Inherited Metabolic Diseases; Lysosomal Storage Disorders; Peroxisomal Storage Diseases; Inborn Errors of Metabolism; Mucopolysaccharidosis
Keywords: Hurler Syndrome; MPS I; Hurler-Scheie Syndrome; Hunter Syndrome; MPS II; Sanfilippo Syndrome; MPS III; Maroteaux-Lamy Syndrome; MPS VI; Krabbe Disease; Globoid Leukodystrophy; Metachromatic Leukodystrophy; MLD; Adrenoleukodystrophy; ALD; Adrenomyeloneuropathy; AMN; Sandhoff Disease; Tay Sachs Disease; Pelizaeus Merzbacher; PMD; Niemann-Pick Disease A; Niemann-Pick Disease B; Alpha-mannosidosis; Inherited metabolic diseases; Inborn errors of metabolism; Lysosomal storage diseases; Peroxisomal storage diseases; Hematopoietic stem cell transplantation; Umbilical cord blood transplantation; Mucopolysaccharidosis; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis III; Mucopolysaccharidosis VI; I Cell disease; Fucosidosis; GM1 Gangliosidosis; Canavan Disease
MeSH Terms: conditions — Lysosomal Storage Diseases; Metabolism, Inborn Errors; Mucopolysaccharidoses; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Sudden Infant Death; Mucopolysaccharidosis III; Mucopolysaccharidosis VI; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Adrenoleukodystrophy; Sandhoff Disease; Tay-Sachs Disease; alpha-Mannosidosis; Mucolipidoses; Fucosidosis; Gangliosidosis, GM1; Canavan Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Biological: ALD-101

INTERVENTIONS:
Biological: ALD-101 — A subpopulation of cord blood cells composed of cells that express a high level of the intracellular enzyme aldehyde dehydrogenase (ALDH).

SUMMARY:
Eligible research subjects will receive an unrelated umbilical cord blood transfusion as a possible cure for their inherited metabolic disease. A portion of cord blood cells (ALD-101) will be separated from the cord blood unit and given approximately 4 hours after the standard cord blood transfusion.

The study will test if the supplemental cells will increase the speed at which normal levels of circulating blood cells are re-established after transplant.

DETAILED DESCRIPTION:
Subjects will be hospitalized and undergo high doses of chemotherapy which will destroy the child's normal cells including their bone marrow (which forms blood cells) in order to prepare their body for the umbilical cord blood transplant. The cord blood transplant is intended to rescue your child's bone marrow from the bad effects of the procedure. The child will receive 80% of a standard cord blood transplant followed by 20% supplemental stem cell called ALD-101.

The study will evaluate if these cells (ALD-101) will repopulate the bone marrow more rapidly after transplant. This would shorten the period of time that the transplanted subject would be at risk for infection and bleeding and would also decrease the number of red blood cell and platelet transfusions needed.

ALD-101 has been used as a supplement to cord blood transplant in twenty-eight children with genetic diseases and malignancy in one previous clinical study that is on-going.

The main purpose of this research study is to test whether a portion of cord blood cells that have been separated from a cord blood unit (ALD-101) will increase the speed at which normal levels of circulating blood cells are re-established after transplant. This is the experimental part of this study. ALD-101 is also being tested to see if it is safe.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of inherited metabolic diseases; including the following:

  * Hurler Syndrome (MPS I)
  * Hurler-Scheie Syndrome
  * Hunter Syndrome (MPS II)
  * Sanfilippo Syndrome A and B(MPS III)
  * Maroteaux-Lamy Syndrome (MPS VI)
  * Krabbe Disease (Globoid Leukodystrophy)
  * Metachromatic Leukodystrophy (MLD)
  * Adrenoleukodystrophy (ALD and AMN)
  * Sandhoff Disease
  * Tay Sachs Disease
  * Pelizaeus Merzbacher (PMD)
  * Niemann-Pick Disease
  * Alpha-mannosidosis
  * I-Cell Disease (ML II)
  * Fucosidosis
  * GM I Gangliosidosis
  * Canavan Disease
* must be <16 years of age at the time of study enrollment
* must have a good performance status (Lansky ≥80%)
* must have adequate function of other organ systems including: kidney, liver, heart and lungs
* must have given valid written informed consent
* must have a minimum life expectancy of at least 6 months
* must be determined to be a good candidate for a standard umbilical cord blood transplant
* must have an IQ >70 or if too young for IQ testing the potential to reach this endpoint by age 5

Exclusion Criteria:

* HIV, Hepatitis B and/or Hepatitis C positive
* concurrently involved in any other clinical study that affects engraftment or immune reconstitution
* uncontrolled seizures, apnea, evidence of aspiration pneumonia, or evidence of brain stem involvement
* uncontrolled infections
* prior allogeneic stem cell transplant with cytoreduction preparative therapy within 12 months of enrollment

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of adjuvant therapy of ALD-101 in accelerating platelet engraftment in patients also receiving a standard unrelated UCBT for treatment of inherited metabolic diseases | 180 Days

SECONDARY OUTCOMES:
To assess the efficacy of ALD-101 in accelerating neutrophil engraftment | 180 Days
To assess the safety of adjuvant therapy of ALD-101 in infusional toxicity, adverse events, and primary graft failure. | 180 Days

CONTACTS AND LOCATIONS:
Overall Officials: James Hinson, MD, Study Director — Aldagen; Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Mt. Sinai Medical Center, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Prasad VK, Kurtzberg J. Emerging trends in transplantation of inherited metabolic diseases. Bone Marrow Transplant. 2008 Jan;41(2):99-108. doi: 10.1038/sj.bmt.1705970. Epub 2008 Jan 7. PMID 18176609
- [Background] Martin PL, Carter SL, Kernan NA, Sahdev I, Wall D, Pietryga D, Wagner JE, Kurtzberg J. Results of the cord blood transplantation study (COBLT): outcomes of unrelated donor umbilical cord blood transplantation in pediatric patients with lysosomal and peroxisomal storage diseases. Biol Blood Marrow Transplant. 2006 Feb;12(2):184-94. doi: 10.1016/j.bbmt.2005.09.016. PMID 16443516
- [Background] Escolar ML, Poe MD, Martin HR, Kurtzberg J. A staging system for infantile Krabbe disease to predict outcome after unrelated umbilical cord blood transplantation. Pediatrics. 2006 Sep;118(3):e879-89. doi: 10.1542/peds.2006-0747. Epub 2006 Aug 21. PMID 16923928
- [Background] Gentry T, Deibert E, Foster SJ, Haley R, Kurtzberg J, Balber AE. Isolation of early hematopoietic cells, including megakaryocyte progenitors, in the ALDH-bright cell population of cryopreserved, banked UC blood. Cytotherapy. 2007;9(6):569-76. doi: 10.1080/14653240701466347. PMID 17882722
- See also: Sponsor's Website — http://www.aldagen.com